CLINICAL TRIAL: NCT06103955
Title: Improving Outcomes in Dysfunctional Breathing Through the Optimization of Muscle Function (OptiMuscle)
Brief Title: OptiMuscle - Improving Respiration by Optimising Muscle Function
Acronym: OptiMuscle
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salford (Other)
Responsible Party: Principal Investigator, Stephen Preece, Professor of Biomechanics and Rehabilitation, University of Salford
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2192
Record Dates: First submitted 2023-10-13; First posted 2023-10-27 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Dysfunctional Breathing; Breathing Pattern Disorder

STUDY DESIGN:
Intervention Model Description: The primary aim is to carry out preliminary testing of the intervention and to use feedback from participants to make small changes to the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Digital Breathing Biofeedback system (Experimental): Patients will receive 4 physiotherapist-guided breathing retraining sessions with the digital breathing biofeedback system.
  Interventions: Behavioral: Digital Breathing Biofeedback system

INTERVENTIONS:
Behavioral: Digital Breathing Biofeedback system — The biofeedback system provides information to the patient and physio about the muscle coordination of breathing.

SUMMARY:
The primary aim will be to understand whether a digital breathing biofeedback system can improve the outcomes of physiotherapist guided breathing retraining.

DETAILED DESCRIPTION:
Approximately 10% of people in the United Kindom exhibit some form of dysfunctional breathing. This term describes a range of conditions which are characterised by an impairment in the muscular control of breathing and which can result in breathlessness, hyperventilation and, in some cases, dizziness. Current clinical assessment techniques and treatments for dysfunctional breathing are low-tech. The investigators propose that patients would get more benefit from a system which uses biofeedback on muscle patterns to guide breathing re-education. The investigators have developed a new digital health system for the clinical management of dysfunctional breathing. The system uses an avatar to provide biofeedback to communicate abnormal muscle function in real-time, guiding patients through a process in which they gradually learn the correct muscular control of breathing. The proposed intervention seeks to understand if the addition of a digital breathing biofeedback system improves the outcomes of physiotherapy guided breathing retraining. Patients awaiting respiratory physiotherapy for dysfunctional breathing will be recruited to receive 4 sessions of breathing retraining with the assistance of the digital breathing biofeedback system. All patients will complete lung function tests and Quality of Life questionnaires pre- and post- treatment. Patients will also be offered an interview to understand their experiences of using the system.

ELIGIBILITY:
Inclusion Criteria:

* Ability to stand and walk independently
* History of breathing difficulties, such as breathlessness and difficult or laboured breathing for at least previous 6 months.
* Clinical diagnosis of dysfunctional breathing, sometimes referred to as breathing pattern disorder.
* If participants have co-existing respiratory problems, e.g. asthma, these should not be felt (in the opinion of the referring clinician) to be the cause of the current symptoms of breathlessness.

Exclusion Criteria:

* Inability to speak and understand English sufficient to read and understand the information sheet and sign the consent form.
* BMI >34
* Currently receiving active treatment for dysfunctional breathing
* Received treatment for acute lower respiratory tract infection or asthma exacerbation with last 4 weeks
* Significant respiratory co-morbidity (i.e. where the major respiratory diagnosis is not asthma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Lung Function | Change from Baseline to 8 weeks
  Spirometry test of lung volume will be measured included tidal volume and forced expiratory volumes. (Larger volumes = better lung function)

SECONDARY OUTCOMES:
Change in Nijmegen Score | Change from Baseline to 8 weeks
  Used to capture the extent of hyperventilation. Score 0-64 (0=no hyperventilation, 64=maximum hyperventilation)
Change in the Brief Illness Perception Questionnaire | Change from Baseline to 8 weeks
  Used ot evaluate cognitive and emotional representations of illness. Score 0-80 (0=no threatening perception of illness, 80=maximum threatening perception of illness)
Change in Patient Health Questionnaire (PHQ-9) | Change from Baseline to 8 weeks
  Used to measure depression.Score 0-28 (0=no depression, 28=maximum depression)
Change in the Generalised anxieity disorder (GAD-7) | Change from Baseline to 8 weeks
  Used to measure anxiety. Score 0-21 (no = no anxieity, 21=maximum anxiety)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Salford, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
The investigators may make the clinical data available through a document which will be linked to the final published journal paper

REFERENCES:
- See also: Related Info — https://hub.salford.ac.uk/human-movement-and-rehabilitation/clinical-rehabilitation/avatar-based-breathing-retraining/